CLINICAL TRIAL: NCT04349527
Title: Comparison of the Cosmetic Results, Quality of Life and Patient Satisfaction Achieved With Round-block and Retroglandular Oncoplastic Breast Conserving Surgeries. Response-adaptive (RAR) Prospective Randomised, Comperative Clinical Study
Brief Title: Comparison of the Cosmetic Results, Quality of Life and Patient Satisfaction Achieved With Round-block and Retroglandular Oncoplastic Breast Conserving Surgeries
Status: Recruiting | Type: Observational
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Dr. Zoltan Matrai, Head of Surgical Oncology, National Institute of Oncology, Hungary
Other Study IDs: RB-vs-RG-BCS
Record Dates: First submitted 2020-04-05; First posted 2020-04-16 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Quality of Life; Patient Satisfaction
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RB Group: In this Group Patients receive round-block oncoplastic breast coserving surgery
  Interventions: Procedure: Round-block Oncoplastic Breast Conserving Surgeries
- RG Group: In this Group Patients receive retrogladular oncoplastic breast coserving surgery
  Interventions: Procedure: Retroglandular Oncoplastic Breast Conserving Surgeries

INTERVENTIONS:
Procedure: Round-block Oncoplastic Breast Conserving Surgeries — We de-epithelize the gap between the double round-lines, and we dissect the dermis from the best localization where we can reach the tumor. If the tumor located close to the skin then we are not performing de-epithelization, we excise it with the skin. We mark every wall of the tumor bed with clips. We dissect the surrounding parenchyma- so called parenchyma pillars- from the pectoral fascia and the skin, and we mobilize it. The line under the skin means, the layer under the subcutis, above the superficial fascia, so gives appropriate blood supply to the skin. After this the incision line should be placed 5 mm from the outer round line, so a dermis pillar should be left, and the skin is dissected from the parenchyma as needed. The outer round line should be tightened with a non-absorbable running Benelli suture to fit the areola then interrupted sutures placed to make tensionless the running intracutaneous suture.
  Groups: RB Group
Procedure: Retroglandular Oncoplastic Breast Conserving Surgeries — We incise the skin slightly lateral in the IMF, around 7 cm long. We dissect with electrocauther the parenchyma with the pectoral fascia from the pectoralis major muscle at least until the mamilla. We incise the fascia along with the parenchyma which contains the tumor and macroscopically 10 mm safe zone. If the tumor is palpable, we turn the parenchyma slightly inside-out, if not, we localize it at the maximum measurement detected according to the ROLL labeling. After marking the tumor bed, we directly adapt the surrounding parenchyma pillars with absorbable sutures, or inverting sutures, or if it requires, we adapt the tumor bed with so-called dual plane mobilization. After revision, we close the fascia with absorbable running suture over the Redon drain then subcutaneous running suture with absorbable suture and finally intracutaneous skin closure.
  Groups: RG Group

SUMMARY:
The aim of this clinical study is to analyze due long term follow-up, the clinical, oncological, aesthetic results and patients' reported quality of life and satisfaction in a responsive-adaptive (RAR) prospective, randomized study at a large number of patients whom receive round-block and retroglandular oncoplastic breast conserving surgeries.

According to the study's hypothesis, breast conserving surgery can be oncologically successful and safe with low complication rates resulting in high rate of patient satisfaction and good quality of life, which can be maintained for a long time after WBI with the application of modern oncoplastic breast conserving surgeries. We assume in this study that against of the earliest and mostly studied round-block oncoplastic surgery, the retroglandular technique, firstly reported in the literature by the current authors, is also adequate for oncologically safe, radical tumor removal that comes with low complication rates, suited for adjuvant treatments and able to offer better cosmetic results (NAC does not distorted, and pathological scar will not develop) than round-block OPS and high rate of patient's satisfaction that can be maintained for long-term.

DETAILED DESCRIPTION:
Introduction In the last four decades of oncological breast surgery, based on Umberto Veronesi and Bernard Fisher's prospective comparative studies, organ conservation became highly significant in the case of early breast cancer with the application of microscopically negative surgical margin and adjuvant whole breast irradiation (WBI), which is proven to offer the same survival chance as mastectomy.[1,2] However, in practice, the apparent benefits of organ conservation shaded by the need of second surgery, 5-30%, (repeated directed re-excision or mastectomy) due to microscopically positive surgical margins; the 3-5 weeks long, logistically demanding radiotherapy; and the cosmetically impaired or distorted breasts that remains almost 30% of the surgeries. [3-5] The latter can be explained by our published previous prospective study that the patients report significantly intolerable cosmetic results after 10% volume loss from the inner quadrants and approximately 15-20% volume loss from the lateral quadrants, when its associates with adjuvant WBI. [6] Aside from volume reduction, during a traditional breast conserving surgery (BCS) the tumor bed is left behind as a cavity, whose posterior wall is composed of the pectoralis major muscle and the pectoral fascia, while its anterior wall is composed of skin. Already in the early postoperative stage, with the removal of the seroma, the skin retracts and adheres to the breast muscles or to the fascia. This process is accelerated by the irreversible of the complete residual parenchyma and the change of the skin's structure, elasticity and microcirculation during WBI. This could result 10-20% shrinkage of the breast. The breast shows a typical deformity with the directly curved incision line above the tumor as a result of secondary wound healing process mentioned above. Compared to the contralateral side its volume shrunk, the nipple dislocated to the axillary fold due to the adhesion of the upper-outer quadrant in case of this quadrant's volume loss and typical bird beak formation occurs in case of lower quadrants' border excision; while a central excision usually results in a so-called doughnut shaped breast with a central retractation. Additional challenge is the reconstruction of the post-BCS breast because it is more complicated and achieves poorer cosmetic results than the post-mastectomy breast construction. [7] In order to prevent the above listed disadvantages of BCS, a sophisticated organ conservation breast-surgery was developed with the adaptation of plastic surgery techniques in the last decade, which was named Oncoplastic Surgery (OPS) by Werner Audretsch. [8] These surgeries are volume reducing breast lift surgeries or their alterations, which are based on the knowledge of breast anatomy - especially on its blood circulation (e.g. Würinger's Septum), and its structural and aesthetic subunits (e.g. inframammary fold (IMF), nipple and areola complex (NAC)). The surgeries require particular plastic surgery knowledge. The OPS based on volume displacement using and mobilizing the glandular pillars to fill the wound cavity using the advantages of breast ptosis, narrowing the overall base diameter and the "footprint", and repositioning the NAC, which left behind after the radical removal of the tumor. The OPS is suitable to perform real quadrantectomy, even with a better aesthetic result then it is preoperatively. According to each segments of the breast, various oncoplastic techniques can be applied, giving the oncoplastic surgeon an unprecedented freedom to offer a personalized solution. The OPSs can be classified based on their technical complexity or on the level of volume (<20% / 20-50%) needed to be replaced (Level I./II.). [9] Following the OPS, the remaining scars caused by radiation become almost invisible, and due to the lack of wound cavity, adhesion does not occur.

The most popular Level I. oncoplastic techniques are the periareolar or round-block techniques, or retroglandular technique, which was first published in the international literature by the current authors. These techniques are for those malignant tumors (cT< 3cm) which could be possibly located centrally in every quadrant and requires wide surgical excision less than 20% of the entire breast. [10, 11] The literature relied on oncoplastic breast conserving techniques is usually limited to retrospective cohort studies, while its prospective randomized comparison with traditional breast conserving surgery cannot be performed due to ethical reasons.

The purpose of the current clinical study is to scientifically analyze and compare the clinical, oncological and aesthetic results of the standardized oncoplastic breast conserving surgical techniques, round-block versus retroglandular, in one center for unilateral, solitary, malignant breast tumors in a responsive-adaptive (RAR) prospective randomized trial with long term follow-up.

Aim of the study The aim of this clinical study is to analyze due long term follow-up, the clinical, oncological, aesthetic results and patients' reported quality of life and satisfaction in a responsive-adaptive (RAR) [12] prospective, randomized study at a large number of patients whom receive round-block and retroglandular oncoplastic breast conserving surgeries.

According to the study's hypothesis, breast conserving surgery can be oncologically successful and safe with low complication rates resulting in high rate of patient satisfaction and good quality of life, which can be maintained for a long time after WBI with the application of modern oncoplastic breast conserving surgeries. We assume in this study that against of the earliest and mostly studied round-block oncoplastic surgery, the retroglandular technique, firstly reported in the literature by the current authors, is also adequate for oncologically safe, radical tumor removal that comes with low complication rates, suited for adjuvant treatments and able to offer better cosmetic results (NAC does not distorted, and pathological scar will not develop) than round-block OPS and high rate of patient's satisfaction that can be maintained for long-term.

Patients and method The participation in this study is voluntary. In this current response-adaptive (RAR) prospective randomized study the applied surgical operations count as routine interventions in the literature, as much as in our Department, with standardized techniques. The applicable round-block and retroglandular oncoplastic breast conserving surgeries do not mean new surgical procedures for the patients, not in their techniques, nor in their indications; the prospective examination serves only as a guarantee for the quantitative and qualitative data collection. The examination does not influence the applied oncological therapies; those are still executed based on the institution's preoperative and postoperative multidisciplinary breast oncological committee's professional decisions.

The study does not change the complex oncological treatment in any ways, considering the NCI protocol.

In this study the response-adaptive classification means that the choice of the optimal surgical procedure for the patient is not influenced by the clinical study. The decision making model is the same as it is in our department, same as for patients that are not participating in the study, so the subgroups chosen according to the oncological morbidity, the location of the tumor (the round-block technique is more appropriate for those ones that are closer to the surface, while the ones located more deeper, closer to the pectoralis major muscle are adequate for the retroglandular procedure), the breast size, the structure and ptosis of parenchyma. The applied and studied surgical techniques like aside of the clinical examination, do not require symmetrization.

The current study does not include intervention in a scientific term due to the above listed reasons, so it is not differs of the routinely used treatment protocol.

The primary endpoint of the study Correlation analysis of oncological control, cosmetic result, patients' satisfaction and quality of life achieved by various surgical techniques; and these follow-ups in one, two, three, four, and five years.

The study's secondary endpoints To determine the complication's ratio of early and late surgeries, and the surgical strain (the length of the surgery and hospitalization).

Based on the results, once it gains scientific confirmation, the retroglandular, oncoplastic breast conserving technique, proposed by the authors for the first time, could become a Level I oncoplastic technique.

Patients:

- Under the age of 65, suffering from unilateral (cT< 3cm) in situ or invasive breast cancer, who are fit for breast conserving surgeries, who had no previous breast surgery, independent from axillary surgery (sentinel lymph node biopsy or axillary block dissection)

Excluding factors:

* In case the patient does not volunteer for the examination or the follow-ups
* Age above 65 years or poor general health condition, where the estimated life expectancies would be less than 2 years even without a tumor
* Malignant invasive tumor in the past history (except for non-melanoma skin tumors)
* Mastectomy performed due to positive resection margin
* Prior breast surgery (e.g. aesthetic surgery, breast lift) and/or radiotherapy on the breast or in the axilla
* Malignant tumor is not removed completely with pathological examination
* Severe non-surgical (e.g. radiotherapy) complication, which could influence the aesthetic and functional results
* Autoimmune diseases
* Tumor requiring mastectomy, or clinically larger than 3 cm tumor primary, or mastitis carcinomatosa, lymphangitis carcinomatosa
* Long-term steroid usage, which changed the skin's quality and structure
* Patient under foster care, or psychically non-cooperative patient

Preoperative examinations:

* Physical examination
* Triplet examination of the breast
* Preoperative core biopsy or FNAB
* Staging examinations: chest x-ray, abdominal ultrasound, bone scintigraphy
* Axillary ultrasound and cytological examination if required
* Required additional imaging based on the oncological staging (targeted x-ray, CT, MRI, PET)
* Routine hematological and blood test analysis
* Measurements of jugulum-nipple width, nipple midline width, and nipple inframammary-fold width
* Measurements of the areola's horizontal and vertical diameter
* Regnault Classification of breasts' ptosis
* Photo documentation (standard 5 directions and ap with raised arms) and the application of the BCCT.core program (regarding data protection regulations) [13]
* Filling out the BREAST-Q questionnaire [14]

Recorded data:

Age, body mass, height, BMI, pre-/postoperative cup sizes, presence of preoperative breast assymetry and its severity (BCCT.core software data), past history, medication, smoking habits, oncological data, cTNM, pTN, pathological data, molecular genetic subtype, neoadjuvant and adjuvant therapy, type of axillary treatment, locoregional cancer recurrance, metastasis.

Postoperative complications were classified following Clavien-Dindo Classification[15, 16] Grade I complication (light inflammations, non-surgical haematoma or suffusion, seroma formation, partial skin/NAC loss, limited fat necrosis, SSI and lymphoedema) does not require medication or surgical treatment. Grade II complication is a Grade I complication that requires medication or surgical interaction (antibiotic therapy, resuture due SSI and multiple puncture due chronic seroma). Grade III complication requires invasive surgical action (haematoma evacuation, chronic inflammation which requires reoperation, severe fat necrosis, full skin/ NAC necrosis and wound dehiscense). Grade IV complication means temporary organ failure. Grade V complication is one that leads to death.

The following data are collected in this trial: preoperative jugulum-nipple width, nipple-midline width, nipple-IMF width, vertical and horizontal width of the areola, Regnault Classification of the breast ptosis then repeating the above measurements during the follow-up (every 6 months) with parallel photo documentation, using BCCT.core program and data recording of the BREAST-Q questionnaire and 5 point Likert-scale.[17]

Methods Enrolled patients who require round-block, or retroglandular oncoplastic breast conserving surgery on one side, they filled out BREAST Q questionnaire and have undergone preoperative photo documentation, BCCT.core software analysis and breast ptosis detection according to Regnault Classification. In case of neoadjuvant therapy, the procedure is the same and the patient selection and data recording are performed preoperatively.

Flow chart

OPS, oncoplastic breast conserving surgery The patients after breast conserving surgery receive adjuvant therapy based on the decision of the multidisciplinary breast cancer board of the Institute. Data collection: measurements of the patients, the photo documentation, filling the BCCT.core software database and the postoperative quality of life BREAST Q questionnaire made postoperatively in the 4th-6th week then in the 3rd postoperative month then after every 6 months. The oncological follow-up carried out by the guideline of the Institute, and the follow-up lasts until the end of the 5th year. During this period, correction of the breast is not allowed.

Surgical therapy The treatment of the patients examined in the study relied on the techniques of the Breast and Sarcoma Department of the National Cancer Institute including standardized round block oncoplastic breast conserving surgery, or the standardized retroglandular oncoplastic technique, which was first described in the literature by our workgroup. (See the detailed description of these: Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019., 10.4. Periareolar oncoplastic technique; 10.13. Retroglandular oncoplastic breast-conserving surgical technique) [18]

The round block oncoplastic breast conserving technique The surgical procedure planned after the exact localization of the cancer in surgical position. In case of non-palpable tumors, the preoperative markings are obligatory (isotope). Considering the previously mentioned facts, we mark in standing position the double round-lines and midline, the footprint and the line between the medioclavicular point and nipple, and its distal extension through the IMF. After desinfection and isolation, we de-epithelize the gap between the double round-lines, and we dissect the dermis from the best localization where we can reach the tumor. We suggest to infiltrate the wound line with adrenaline diluted saline (1:1000) before the incision to avoid the continuous bleeding of the subdermal plexus, which can disturb the procedure. If the tumor located close to the skin then we are not performing de-epithelization, we excise it with the skin. We mark every wall of the tumor bed with clips. After oncologically safe resection (resection border, tumor bed marking, intraoperative specimen mammography/ultrasound and control of the pathological "safe border" macroscopically), we dissect the surrounding parenchyma- so called parenchyma pillars- from the pectoral fascia and the skin, and we mobilize it. The line under the skin means, the layer under the subcutis, above the superficial fascia, so gives appropriate blood supply to the skin. The mobilization of the parenchyma pillars should be done adequately with absorbable sutures to avoid dead space, skin intrusion and breast deformity. After this the incision line should be placed 5 mm from the outer round line, so a dermis pillar should be left, and the skin is dissected from the parenchyma as needed. The outer round line should be tightened with a non-absorbable running Benelli suture to fit the areola then interrupted sutures placed to make tensionless the running intracutaneous suture. A subcutaneous drain should be left if needed until the 2nd postoperative day. We use a slight compression bandage for 12 hours. The wound should be covered according to the general surgical rules, if possible, using Steri-strip (topical mupirocin cream suggested on it), the sutures removed after 2-3 weeks.

The retroglandular oncoplastic breast conserving technique We mark the midline and the breast's footprint in standing position. After desinfection and isolation in the OR, we infiltrate the subdermal plexus with the above mentioned way then we incise the skin slightly lateral in the IMF, around 7 cm long. We dissect with electrocauther the parenchyma with the pectoral fascia from the pectoralis major muscle at least until the mamilla. If the tumor's localization requires until the whole footprint is reached. We incise the fascia along with the parenchyma which contains the tumor and macroscopically 10 mm safe zone. If the tumor is palpable, we turn the parenchyma slightly inside-out, if not, we localize it at the maximum measurement detected according to the ROLL labeling. We mark the specimen and then send it to pathological examination, if needed intraoperative mammography and/or hystological examination. After marking the tumor bed, we directly adapt the surrounding parenchyma pillars with absorbable sutures, or inverting sutures, or if it requires, we adapt the tumor bed with so-called dual plane mobilization. The sentinel lymph node biopsy is performed from the same incision, while in case of axillary dissection, we perform it in a separate ca. 6 cm long incision line placed in the axillary fold. After revision, we close the fascia with absorbable running suture over the Redon drain then subcutaneous running suture with absorbable suture and finally intracutaneous skin closure. The Redon planned to be removed 50 ml/day.

The surgery required localization technique of the Institute, in case of non-palpable cancer, is the routinely used ultrasound guided or stereotaxic isotope labeling technique (ROLL), which marker is the same as the radiolabeled 99Tc albumin solution in sentinel lymph node biopsy.

According to the valid protocol of the National Cancer Institute, the surgery of the axilla can be either sentinel lymph node biopsy or axillary lymphadenectomy/ axillary block dissection, if needed with radiotherapy of the axillary and supraclavicular region depending on the regional stage of the breast cancer. (see as well in Z Mátrai, G Gulyás, T Kovács, M Kásler Principles and practice of oncoplastic breast surgery. Medicina Kiadó Zrt, 2019. 8. fejezet: Tradicional breast surgery, 8.1.2. Axillary lymph nodee dissection; 9. Sentinel lymph node biopsy in breast cancer)[18]

Using and collecting cosmetic results The following data collected in standing position marking the midline and the IMF preoperatively then postoperatively in the 4th-6th week then in the 3rd postoperative month then after every 6 months: jugulum-nipple width, nipple-midline width, horizontal and vertical width of the areola and nipple-IMF width The breast ptosis examination performed according to Regnault Classification at the beginning and after symmetrization.

The primary aesthetic stage will be documented with standard photo documentation using valid BCCT.core software making it measurable which allows us to compare it. the photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. The patients are anonymous on the pictures without their faces, and the photo documentation performed without jewelry. The mentioned software counts measurements regarding to the photo documentation and gives a 4-point rating scale (1: excellent, 2: good, 3: acceptable, 4: non-acceptable). These numerical results can be statistically analyzed.

The quality of life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "satisfaction with the breast", "discomfort by radiotherapy", "psychosexual wellbeing" and "physical wellbeing". We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better quality of life. [14] The questionnaires are filled before the procedure and after the surgery 4th-6th weeks then postoperatively in the 3rd months and every 6th months.

We use the Likert scale (1. definitely not, 2: no, 3: abstain, 4: agree, 4: definitely agree) for evaluating the subjective aesthetic outcome based on the photo documentation (preoperative, postoperative 4-6th weeks, 3rd months, every 6 months 5 years long). Based on the photo documentation three, non-involved breast surgeons make the evaluation separately without communication. The results are collected and averaged.

Follow-up The follow-up is similar to the surgical and oncological follow-up in the National Cancer Institute, so it is not a burden for the patients The primary check-up and data registration performed preoperatively, the second check-up performed 4-6th weeks after the oncoplastic procedure then 3rd postoperative months with photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire.

After this the photo documentation, body measurements, body mass calculation and BREAST-Q questionnaire examination performed every 6 months until the 5th year.

The bioethical background of the study It is a non-interventional clinical study is conducted by the competent regional research ethics committees in accordance with the Medical law 164 / A. § (2).

This non-interventional clinical trial is performed with the permission of the Ethical Committee of the National Cancer Institute according to the 23/2002. (V.9.) Medical Regulation.

The Researchers commit themselves to protect the patient's data, photo documentation in accordance with the WHO Good Clinical Practice ( based on the Helsinki Declaration) and the applicable provisions of the General Data Protection Regulation (GDPR) regarding the international ethical and scientific quality requirements pertaining to the design, conduct, documentation and reporting principles of tests conducted on humans.

Data collection and registration It is performed with the registration sheet for computer processing and BREAST-Q questionnaire which is an internationally validated and authorized mirror translated questionnaire. Digital photo documentation (standard 5 direction with lowered arms and ap direction with raised arms) The BCCT.core made with at least 9 megapixel photo documentation, ap and lateral directions with lowered and raised arm to calculate numerically with a validated procedure the aesthetic outcome.

Planned number of patients The planned number of the patients(calculated patients number plus 10%): 110x2=220+ 22 cases ∑242 cases should be included.

Planned time of patient inclusion: 1 year. Planned follow-up time The planned follow-up time after reconstruction and symmetrization is 5 year. Interim analysis performed after 2 years median follow-up period. Final analysis is performed 5 years after closing the patient inclusion period.

ELIGIBILITY:
Inclusion Criteria:

* - Under the age of 65, suffering from unilateral (cT< 3cm) in situ or invasive breast cancer, who are fit for breast conserving surgeries, who had no previous breast surgery, independent from axillary surgery (sentinel lymph node biopsy or axillary block dissection)

Exclusion Criteria:

* In case the patient does not volunteer for the examination or the follow-ups
* Age above 65 years or poor general health condition, where the estimated life expectancies would be less than 2 years even without a tumor
* Malignant invasive tumor in the past history (except for non-melanoma skin tumors)
* Mastectomy performed due to positive resection margin
* Prior breast surgery (e.g. aesthetic surgery, breast lift) and/or radiotherapy on the breast or in the axilla
* Malignant tumor is not removed completely with pathological examination
* Severe non-surgical (e.g. radiotherapy) complication, which could influence the aesthetic and functional results
* Autoimmune diseases
* Tumor requiring mastectomy, or clinically larger than 3 cm tumor primary, or mastitis carcinomatosa, lymphangitis carcinomatosa
* Long-term steroid usage, which changed the skin's quality and structure
* Patient under foster care, or psychically non-cooperative patient

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The aim of the clinical study is to measure with a long-term follow-up and with qualitative and quantitative indicators the changes in cosmetic results, quality of life and patient satisfaction after delayed- immediate breast reconstruction with standardized technique Skin Reducing Nipple sparing mastectomy, SRNSM and SSM. The planned subgroups contain 50-50 cases. Planned number of patients (calculated patients' number plus 10%): 50x2=100 +10 cases
  * 110 cases should be included.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2020-04-18 (Actual); Primary Completion 2022-04-05 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
Oncological safety | five years follow up
  Correlation analysis of oncological control (overall and disease free survival) achieved by various surgical techniques. The follow-up is similar to the surgical and oncological follow-up in the National Cancer Institute, so it is not a burden for the patients. The overall and disease free survival is calculated from the surgigal treatment to first event. The event such as death, local recurrence, locoregional recurrence or distant metasasis will be recorded.
Cosmetic results | five years follow up
  The primary aesthetic stage will be documented with standard photo documentation using valid BCCT.core software making it measurable which allows us to compare it. the photo documentation performed the standard way in 5 position (antero-posterior (ap), 45 degree oblique and 90 degree lateral), in ap direction both ways arms up and down with strict adherence to personal privacy policies. The mentioned software counts measurements regarding to the photo documentation and gives a 4-point rating scale (1: excellent, 2: good, 3: acceptable, 4: non-acceptable). These numerical results can be statistically analyzed. We use the Likert scale (1. definitely not, 2: no, 3: abstain, 4: agree, 4: definitely agree) for evaluating the subjective aesthetic outcome based on the photo documentation (preoperative, postoperative 4-6th weeks, 3rd months, every 6 months 5 years long). The results are collected and averaged.
Patients' satisfaction | five years follow up
  Correlation analysis of patients' satisfaction achieved by various surgical techniques. The patients' satisfaction life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "satisfaction with the breast", "discomfort by radiotherapy" We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better patients' satisfaction. The questionnaires are filled before the procedure and after the surgery 4th-6th weeks then postoperatively in the 3rd months and every 6th months.
Quality of life | five years follow up
  Correlation analysis of quality of life achieved by various surgical techniques. The quality of life is measured by BREAST-Q validated questionnaire. According to this, we give a score in a 1-100 scale measuring the variables of "psychosexual wellbeing" and "physical wellbeing". We use preoperatively a preoperative questionnaire and postoperatively a postoperative questionnaire. Higher rates show better quality of life. The questionnaires are filled before the procedure and after the surgery 4th-6th weeks then postoperatively in the 3rd months and every 6th months.

SECONDARY OUTCOMES:
Complication's ratio | 5 years follow up
  Postoperative complications were classified following Clavien-Dindo Classification. Grade I complication (light inflammations, non-surgical haematoma or suffusion, seroma formation, partial skin/NAC loss, limited fat necrosis, SSI and lymphoedema) does not require medication or surgical treatment. Grade II complication is a Grade I complication that requires medication or surgical interaction (antibiotic therapy, resuture due SSI and multiple puncture due chronic seroma). Grade III complication requires invasive surgical action (haematoma evacuation, chronic inflammation which requires reoperation, severe fat necrosis, full skin/ NAC necrosis and wound dehiscense). Grade IV complication means temporary organ failure. Grade V complication is one that leads to death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Singletary SE. Surgical margins in patients with early-stage breast cancer treated with breast conservation therapy. Am J Surg. 2002 Nov;184(5):383-93. doi: 10.1016/s0002-9610(02)01012-7. PMID 12433599
- [Background] Cochrane RA, Valasiadou P, Wilson AR, Al-Ghazal SK, Macmillan RD. Cosmesis and satisfaction after breast-conserving surgery correlates with the percentage of breast volume excised. Br J Surg. 2003 Dec;90(12):1505-9. doi: 10.1002/bjs.4344. PMID 14648728
- [Background] Matrai Z, Gulyas G, Toth L, Polgar C, Bidlek M, Szabo E, Lang I, Horvath Z, Udvarhelyi N, Kunos C, Savolt A, Pesthy P, Kasler M. [Challenges in oncologic plastic surgery of the breast]. Magy Onkol. 2011 Mar;55(1):40-52. Epub 2011 Mar 31. Hungarian. PMID 21617790
- [Background] Pukancsik D, Kelemen P, Ujhelyi M, Kovacs E, Udvarhelyi N, Meszaros N, Kenessey I, Kovacs T, Kasler M, Matrai Z. Objective decision making between conventional and oncoplastic breast-conserving surgery or mastectomy: An aesthetic and functional prospective cohort study. Eur J Surg Oncol. 2017 Feb;43(2):303-310. doi: 10.1016/j.ejso.2016.11.010. Epub 2016 Dec 5. PMID 28069398
- [Background] Hamdi M. Oncoplastic and reconstructive surgery of the breast. Breast. 2013 Aug;22 Suppl 2:S100-5. doi: 10.1016/j.breast.2013.07.019. PMID 24074768
- [Background] Audretsch W. [Space-holding technic and immediate reconstruction of the female breast following subcutaneous and modified radical mastectomy]. Arch Gynecol Obstet. 1987;241 Suppl:S11-9. doi: 10.1007/BF00930983. No abstract available. German. PMID 3426257
- [Background] Clough KB, Kaufman GJ, Nos C, Buccimazza I, Sarfati IM. Improving breast cancer surgery: a classification and quadrant per quadrant atlas for oncoplastic surgery. Ann Surg Oncol. 2010 May;17(5):1375-91. doi: 10.1245/s10434-009-0792-y. Epub 2010 Feb 6. PMID 20140531
- [Background] Matrai Z, Ujhelyi M, Kovacs T, Kelemen P, Savolt A, Kovacs E, Eles K, Meszaros N, Kenessey I, Stamatiou A, Pukancsik D. Evaluation of a Retroglandular Oncoplastic Technique as a Standard Level I Oncoplastic Breast-Conserving Surgery: A Retrospective Clinicopathologic Study of 102 Patients With Breast Cancer. Clin Breast Cancer. 2019 Jun;19(3):e459-e467. doi: 10.1016/j.clbc.2019.02.005. Epub 2019 Feb 20. PMID 30992191
- [Background] Benelli L. A new periareolar mammaplasty: the "round block" technique. Aesthetic Plast Surg. 1990 Spring;14(2):93-100. doi: 10.1007/BF01578332. PMID 2185619
- [Background] Rosenberger WF, Sverdlov O, Hu F. Adaptive randomization for clinical trials. J Biopharm Stat. 2012;22(4):719-36. doi: 10.1080/10543406.2012.676535. PMID 22651111
- [Background] Cardoso JS, Cardoso MJ. Towards an intelligent medical system for the aesthetic evaluation of breast cancer conservative treatment. Artif Intell Med. 2007 Jun;40(2):115-26. doi: 10.1016/j.artmed.2007.02.007. Epub 2007 Apr 8. PMID 17420117
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Dikmans REG, Nene LEH, Bouman MB, de Vet HCW, Mureau MAM, Buncamper ME, Winters HAH, Ritt MJPF, Mullender MG. The Aesthetic Items Scale: A Tool for the Evaluation of Aesthetic Outcome after Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Mar 1;5(3):e1254. doi: 10.1097/GOX.0000000000001254. eCollection 2017 Mar. PMID 28458968
- [Background] Mátrai Z GG, Kovács T, Kásler M Principles and practice of oncoplastic breast surgery. Medicina Kiadó; 2019.